CLINICAL TRIAL: NCT02303171
Title: Use of Warfarin After the First Trimester in Pregnant Women With Antiphospholipid Syndrome
Brief Title: Use of Warfarin After the First Trimester in Pregnant Women With APS
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mohamed Sayed Abdelhafez (Other)
Responsible Party: Sponsor-Investigator, Mohamed Sayed Abdelhafez, Dr, Mansoura University
Organization: Mansoura University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MIE1
Record Dates: First submitted 2014-11-25; First posted 2014-11-27 (Estimated); Last update posted 2023-10-31 (Actual); Status verified 2023-10

CONDITIONS: Recurrent Miscarriage; Antiphospholipid Syndrome
Keywords: Antiphospholipid syndrome; APS; Warfarin
MeSH Terms: conditions — Abortion, Habitual; Antiphospholipid Syndrome | interventions — Enoxaparin; Warfarin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Enoxaparin group (Active Comparator): Women will be subjected to anticoagulant therapy by Enoxaparin throughout pregnancy
  Interventions: Drug: Enoxaparin
- Warfarin group (Active Comparator): Women will be subjected to anticoagulant therapy by Enoxaparin in the first trimester then Warfarin after the first trimester
  Interventions: Drug: Warfarin

INTERVENTIONS:
Drug: Enoxaparin — Women will be given Enoxaparin throughout pregnancy in a dose of 40 mg/day subcutaneously (SC)
  Other Names: Clexan
  Arms: Enoxaparin group
Drug: Warfarin — Women will be given Enoxaparin (40 mg/day SC) in the first trimester then Warfarin (3-5 mg/day) after the first trimester until termination of pregnancy
  Other Names: Marevan
  Arms: Warfarin group

SUMMARY:
Evaluation of shifting to oral vitamin K antagonist after the first trimester instead of using low molecular weight heparin (LMWH) throughout pregnancy in pregnant women with antiphospholipid syndrome (APS)

DETAILED DESCRIPTION:
Women will be randomly divided into two groups; one will be subjected to anticoagulant therapy by Enoxaparin throughout pregnancy and the other will be subjected to anticoagulant therapy by Enoxaparin in the first trimester then Warfarin after the first trimester until termination of pregnancy.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women with APS diagnosed according to the revised classification criteria for APS in 2006 in Sydney, Australia
* Early pregnancy body weight is 50-90 Kg

Exclusion Criteria:

* Women with systemic lupus erythematosus (SLE)
* Women with active thromboembolic disorders
* Women with history of previous thromboembolic disorders

Ages: 20 Years to 38 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2014-11; Primary Completion 2024-12 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Fetal loss | From 12 weeks to 42 weeks gestational age
  Unexplained fetal death of morphologically normal fetus after the first trimester

SECONDARY OUTCOMES:
Preterm delivery | From 20 weeks to 34 weeks gestational age
  Delivery of morphologically normal fetus before 34 weeks of gestation due to severe preeclampsia or placental insufficiency
Intrauterine growth restriction (IUGR) | At birth
  Birth weight less than the 10th percentile for gestational age
Congenital fetal malformations | At birth
  Congenital fetal malformations

OTHER OUTCOMES:
Hemorrhagic complications | After 12 weeks gestational age up to birth
  Hemorrhagic complications
Thromboembolic complications | After 12 weeks gestational age up to birth
  Thromboembolic complications

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed I Eid, Dr, Principal Investigator — Mansoura University; Mohamed S Abdelhafez, Dr, Study Director — Mansoura University; Abdelmageed F Mashaly, Prof, Study Chair — Mansoura University
Locations (2):
- Egypt (2):
  - Obstetrics and Gynecology Department in Mansoura University Hospital, Al Mansurah, Dakahlia Governorate
  - Private practice settings, Al Mansurah, Dakahlia Governorate

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hamulyak EN, Scheres LJ, Marijnen MC, Goddijn M, Middeldorp S. Aspirin or heparin or both for improving pregnancy outcomes in women with persistent antiphospholipid antibodies and recurrent pregnancy loss. Cochrane Database Syst Rev. 2020 May 2;5(5):CD012852. doi: 10.1002/14651858.CD012852.pub2. PMID 32358837